CLINICAL TRIAL: NCT01536041
Title: A Double-blind, Placebo-controlled, Four-way Crossover Study to Compare the Safety and Efficacy of ONO-6950 20 mg and 200 mg QD Versus Placebo and Montelukast (Singulair) in Asthmatic Patients Who Experience Exercise-induced Bronchoconstriction
Brief Title: A Placebo and Active Controlled Study of ONO-6950 in Asthmatic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-6950POU006
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
Keywords: asthma; Adult
MeSH Terms: conditions — Asthma | interventions — gemilukast; montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Experimental 200 mg dose (Experimental)
  Interventions: Drug: ONO-6950
- Experimental 20 mg dose (Experimental)
  Interventions: Drug: ONO-6950
- Active Comparator Montelukast (Active Comparator)
  Interventions: Drug: Montelukast
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-6950 — 200 mg QD, single dose
  Arms: Experimental 200 mg dose
Drug: ONO-6950 — 20 mg QD, single dose
  Arms: Experimental 20 mg dose
Drug: Montelukast — 10 mg Montelukast, QD single dose
  Arms: Active Comparator Montelukast
Drug: Placebo — Placebo to match ONO-6950 tablets or leukotriene receptor antagonist (LTRA) tablets dosed in a similar manner
  Arms: Placebo Comparator

SUMMARY:
The primary objectives of this study are:

i. to determine the effect of single oral doses (20 and 200 mg) of ONO-6950 versus placebo on exercise induced bronchoconstriction (EIB) as percent attenuation in the decrease of forced expiratory volume in 1 second (FEV1) after exercise challenge

ii. to determine the safety and tolerability of single dose administrations of 20 and 200 mg of ONO-6950 in asthmatic patients.

The secondary objectives of this study are:

i. to compare the effect of different (20 and 200 mg) single oral doses of ONO-6950 versus montelukast (10 mg) on EIB as percent attenuation in the decrease of FEV1 after exercise challenge

ii. to determine the ratio of responders/non-responders in FEV1 for different (20 and 200 mg) single oral doses of ONO-6950 in comparison to montelukast (10 mg) and placebo.

DETAILED DESCRIPTION:
The study will examine if ONO-6950 could alleviate EIB in asthmatic patients. Eligible patients will complete a randomized, double-blind, four-way crossover study. During each of four evaluation periods, patients will be administered a single dose of either 20 or 200 mg ONO-6950, 10 mg Montelukast, or placebo. Each evaluation period include various assessments following exercise challenge in an ambulatory setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders, between 18 to 60 years of age, with bronchial asthma for at least 6 months and history of exercise induced bronchospasm
* Patients with FEV1 ≥ 70% of predicted after withholding short-acting β agonists for at least 8 hours prior to testing
* Screening exercise challenge demonstrates that the patient experiences a fall in FEV1 of ≥ 20%
* Non-smokers with free from the usage of nicotine-containing products at least for a year prior to screening

Exclusion Criteria:

* Previous history of life-threatening asthma, respiratory tract infection and/or exacerbation of asthma within 6 weeks prior to the first screening visit
* History of being unable to tolerate or complete an exercise challenge and clinically significant multiple drug or food allergies
* Past or present disorders and diseases including, but are not limited to cardiovascular, malignancy, hepatic, renal, hematological, neurological, psychiatric, endocrine, or pulmonary other than asthma
* Patients with Seasonal Allergic Rhinitis (SAR) or seasonal allergic asthma,with significant symptoms that may confound study assessment
* Significant safety laboratory, ECG, or vital sign abnormalities that would place the patient at undue risk during the study procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Inhibition of maximum fall in Forced Expiratory Volume in One Second (FEV1) after exercise | 60 minutes following the exercise challenge

SECONDARY OUTCOMES:
AUC (0-30 min) | 30 minutes following the exercise challenge
  area under the concentration time curve integrating fall in FEV1 following exercise over the 30 minute interval immediately following exercise
AUC (0-60 min) | 60 minutes following the exercise challenge
  area under the concentration time curve integrating fall in FEV1 following exercise over the 60 minute interval immediately following exercise
Time to recovery of FEV1 to within 5% of the pre-exercise baseline | 90 minutes following the exercise challenge
Proportion of patients using a short acting beta agonist (rescue medication) | 90 minutes following the exercise challenge
Ratio of responder/non-responder in FEV1 | 60 minutes following the exercise challenge

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (9):
- United States (9):
  - Los Angeles Clinical Site 110, Los Angeles, California
  - San Diego Clinical Site 140, San Diego, California
  - Denver Clinical Site 160, Denver, Colorado
  - North Dartmouth Clincial Site 150, North Dartmouth, Massachusetts
  - Minneapolis Clinical Site 190, Minneapolis, Minnesota
  - Princeton Clinical Site 170, Princeton, New Jersey
  - Raleigh Clinical Site 130, Raleigh, North Carolina
  - New Braunfeis Clinical Site 120, New Braunfels, Texas
  - San Antonio Clinical Site 180, San Antonio, Texas